CLINICAL TRIAL: NCT07107958
Title: Assessment of Tongue Diagnosis Changes Before and After Electroacupuncture in Early Rehabilitation of Ischemic Stroke Patients Using ZMT-1A Tongue Analysis System
Brief Title: Electroacupuncture-Induced Changes in Tongue Features in Early Stroke Patients Using ZMT-1A Imaging System
Acronym: ZMT-StrokeEA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Nguyen Ngo Le Minh Anh MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr Nguyen Ngo Le Minh Anh MD, PhD, Lecturer, Faculty of Traditional Medicine, University of Science Ho Chi Minh City
Organization: University of Science Ho Chi Minh City (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZMT-StokeEA2025
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Ischemia Stroke; Electro-acupuncture
Keywords: Electroacupuncture,; Ischemic Stroke; Stroke Rehabilitation; Tongue Diagnosis; ZMT-1A; Barthel Index
MeSH Terms: conditions — Ischemic Stroke | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: This is a single-arm, pre-post interventional study evaluating the effect of electroacupuncture on tongue features and functional outcomes in ischemic stroke patients.
Masking Description: Not applicable. This study is open-label and does not involve blinding of participants or assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electroacupuncture for Ischemic Stroke Rehabilitation (Experimental): Participants with ischemic stroke in the early recovery stage (day 2 to 3 months post-onset) will receive a standardized 4-week course of electroacupuncture, using acupoints based on national clinical guidelines. Electroacupuncture is performed 1 session per day, 5 days per week, targeting acupoints such as LI15 (Jianyu), LI11 (Quchi), TE5 (Waiguan), LI4 (Hegu), GB30 (Huantiao), ST36 (Zusanli), and GB34 (Yanglingquan).
  Tongue images will be collected using the ZMT-1A Tongue Imaging System before and after the intervention. Functional outcomes will be assessed using the Barthel Index
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Electroacupuncture is applied using standardized stroke rehabilitation protocols. Needles are inserted at acupoints including LI15 (Jianyu), LI11 (Quchi), TE5 (Waiguan), LI4 (Hegu), GB30 (Huantiao), ST36 (Zusanli), and GB34 (Yanglingquan), and connected to an electroacupuncture device delivering alternating current stimulation at 10-20 Hz. Each session lasts 15-20 minutes, performed once daily, 5 days per week, for 4 weeks. The intervention follows Vietnam's national traditional medicine guidelines for post-stroke recovery.

SUMMARY:
This prospective clinical study aims to evaluate changes in tongue characteristics before and after a four-week course of electroacupuncture in patients undergoing early rehabilitation following ischemic stroke. Electroacupuncture is widely used in Vietnam as part of traditional medicine-based stroke rehabilitation, yet few studies have objectively quantified its effects on tongue diagnosis.

The study uses the ZMT-1A Tongue Imaging System, an automated diagnostic tool developed in China and currently used at the University of Medicine and Pharmacy at Ho Chi Minh City. The system enables standardized tongue image acquisition and analysis of key features such as tongue body color, tongue shape, coating color, and coating texture.

A total of 385 participants with confirmed ischemic stroke in the early recovery stage (from day 2 to 3 months post-stroke) will be recruited from three hospitals. Each participant will receive electroacupuncture treatment according to standardized protocols for 4 weeks. Tongue images will be collected before and after the intervention. The primary outcome is the change in tongue characteristics. Secondary outcomes include changes in functional status as measured by the Barthel Index and the correlation between tongue changes and functional improvement.

This study aims to provide evidence for the clinical relevance of tongue diagnosis in stroke rehabilitation and to explore its role in monitoring treatment response to electroacupuncture.

DETAILED DESCRIPTION:
Tongue diagnosis is one of the four traditional diagnostic methods in Chinese and Vietnamese traditional medicine. It reflects the physiological and pathological conditions of the internal organs and is considered an objective and noninvasive indicator for syndrome differentiation. However, tongue diagnosis has historically relied on practitioner experience, which may be subject to environmental conditions and inter-observer variability.

In recent years, automated tongue diagnostic systems (ATDS) have been developed to standardize and objectify tongue assessment. One such system, ZMT-1A, is equipped with a controlled lighting environment, a calibrated camera, and built-in algorithms for analyzing tongue body and coating features. This study uses the ZMT-1A system to capture and analyze tongue images of stroke patients undergoing electroacupuncture treatment.

Ischemic stroke is a leading cause of long-term disability worldwide. Early rehabilitation within the first 3 months post-stroke is essential for functional recovery. In Vietnam, electroacupuncture is integrated into standard care for stroke rehabilitation and is believed to regulate qi and blood, restore meridian circulation, and support organ function. Yet, few studies have examined the effects of electroacupuncture on tongue characteristics, which may reflect internal changes and treatment response.

This single-group pre-post interventional study will recruit 385 patients diagnosed with ischemic stroke in the early recovery stage (day 2 to 3 months post-onset) from three clinical sites: the Ho Chi Minh City Hospital for Rehabilitation and Orthopedics, the Ho Chi Minh City Traditional Medicine Hospital, and University Medical Center - Campus 3. All participants will receive a 4-week course of electroacupuncture based on national standardized acupoint protocols for stroke.

Data collection will include: (1) tongue images before and after treatment, captured using the ZMT-1A system; and (2) functional assessment using the Barthel Index. The main outcome measure is the change in tongue characteristics, specifically tongue body color, shape, coating color, and coating texture. Secondary outcomes include improvement in Barthel Index score and correlation between tongue features and functional recovery.

The study was approved by the Ethics Committee in Biomedical Research at the University of Medicine and Pharmacy at Ho Chi Minh City (Approval No. 2862/ĐHYD-HĐĐĐ, dated October 10, 2024). The findings of this study may support the clinical validity of tongue diagnosis and promote the use of image-based diagnostic systems in traditional medicine research and practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults of any age (no upper or lower age limit).
* Diagnosis of ischemic stroke confirmed by neuroimaging (CT or MRI).
* Currently in the early recovery phase, defined as 2 days to 3 months after stroke onset.
* Stable vital signs and deemed clinically suitable for rehabilitation and electroacupuncture.
* Ability to communicate effectively and follow treatment instructions.
* Provides written informed consent to participate in the study.

Exclusion Criteria:

* Diagnosis of hemorrhagic stroke or stroke of non-ischemic origin.
* Severe cognitive deficits or global aphasia that prevents participation or assessment.
* Serious comorbid conditions such as end-stage heart failure, malignancies, or renal failure.
* Presence of electronic implants (e.g., pacemakers) or other contraindications to electroacupuncture.
* Enrollment in another interventional clinical trial within the preceding 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Change in tongue diagnosis characteristics before and after electroacupuncture treatment | Baseline and after 4 weeks of electroacupuncture
  This outcome assesses the changes in tongue features including:
  * Tongue body color
  * Tongue shape
  * Tongue coating color
  * Tongue coating texture
  Images are captured pre- and post-electroacupuncture using the ZMT-1A Tongue Imaging System. The system automatically classifies tongue features into standardized categories (25-parameter classification system).
  Unit of Measure:
  Proportion (%) of participants showing improvement or change in each tongue characteristic (ordinal scale)

SECONDARY OUTCOMES:
Change in Barthel Index score before and after electroacupuncture treatment | Baseline and after 4 weeks of electroacupuncture
  This outcome evaluates the change in functional independence using the Barthel Index, a validated 10-item scale assessing activities of daily living (ADLs). Scores range from 0 (completely dependent) to 100 (fully independent).
  Unit of Measure:
  Mean Barthel Index score (scale: 0-100)

OTHER OUTCOMES:
Correlation between changes in tongue features and changes in Barthel Index score | Baseline and after 4 weeks of electroacupuncture
  This outcome measures the statistical correlation between:
  * The degree of change in tongue characteristics (ordinal scores based on ZMT-1A analysis)
  * The improvement in Barthel Index score
  * The strength of association will be evaluated using Pearson or Spearman correlation coefficients, depending on data distribution.
  Unit of Measure:
  Correlation coefficient (r-value), p-value

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Anh Nguyen Ngo Le, M.D., Ph.D., Principal Investigator — Faculty of Traditional Medicine, UMP, HCMC
Locations (3):
- Vietnam (3):
  - Ho Chi Minh City Traditional Medicine Hospital, Ho Chi Minh City
  - University Medical Center Ho Chi Minh City - Campus 3, Ho Chi Minh City
  - Ho Chi Minh City Hospital for Rehabilitation and Orthopedics, Ho Chi Minh City